CLINICAL TRIAL: NCT05618522
Title: Clinical Outcomes of Low Temperature Vacuum-dehydrated Amnion Membrane (Omnigen) in Treatment of Acute Chemical Eye Injuries
Brief Title: Omnigen in Acute Chemical Eye Injuries
Acronym: Omnigen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Nancy Maher, Senior regsistrarof ophthalmology, Farwaniya Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Omnigen; associate professor (Registry Identifier: Nancy Maher)
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Acute Chemical Eye Injuries
Keywords: amniotic membrane; chemical eye injury

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the lens loaded with Omnigen (Other): patients with acute chemical eye injury treated with omnigen
  Interventions: Procedure: vacuum-dehydrated amnion membrane (omnigen); Device: the lens loaded with Omnigen

INTERVENTIONS:
Procedure: vacuum-dehydrated amnion membrane (omnigen) — applying the lens loaded with Omnigen on the cornea
  Other Names: application of amnilenz
Device: the lens loaded with Omnigen — the lens loaded with Omnigen

SUMMARY:
evaluation of the role of Omnigen in acute chemical eye injuries

DETAILED DESCRIPTION:
prospective interventional study included patients with different degrees of acute chemical eye injuries were treated by Omnigen and followed up for one month

ELIGIBILITY:
Inclusion Criteria:

* acute chemical eye injury

Exclusion Criteria:

* absent or shallow fornices
* symblepharon interfering with lens placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Epithelial healing | 1 week
  slit lamp examination with cobalt blue light after installing fluroscein drops
limbal ischaemia | 1 week
  slit lamp examination of the clock hours of vascularity around the limbususing both Due classification and Roper Hall

SECONDARY OUTCOMES:
omnigen tolerability | 1 week
  questionnaire for the patients asking about discomfort sensation or the need to patch the eye

CONTACTS AND LOCATIONS:
Locations (1):
- Farwanyia Hospital, Al Farwānīyah, Farwanyia, Kuwait

IPD SHARING:
Plan to Share IPD: No